CLINICAL TRIAL: NCT04719390
Title: BabySTEPs: Supportive Texts to Empower Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The National Center on Addiction and Substance Abuse at Columbia University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BabySTEPs; R34AA028407 (NIH)
Record Dates: First submitted 2020-12-09; First posted 2021-01-22 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Drinking
Keywords: Text messaging
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Micro-Randomized Trial (MRT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Text Messaging Intervention (Experimental): After each daily EMA survey, participants were micro-randomized to (1) receive a maternal-focused message (.40 probability); (2) receive a drinking-focused message (.40 probability) or (3) receive no message (.20 probability).
  Interventions: Behavioral: Text Message

INTERVENTIONS:
Behavioral: Text Message — Maternal-Focused Message: When randomized to receive a maternal-focused message, participants will receive a message that is focused on the transition to motherhood and the joys and challenges of caring for a newborn.
  Drinking-Focused Message:
  When randomized to receive a drinking-focused message, participants will receive a message that is focused on reducing alcohol use.
  All messages of both types are designed to map onto behavior change techniques that are empirically supported for alcohol use.

SUMMARY:
This study is a pilot micro-randomized trial (MRT) that aims to establish feasibility, acceptability, and preliminary proof-of-concept of a text messaging intervention for postpartum alcohol use.

DETAILED DESCRIPTION:
The pilot MRT is designed preliminary to assess feasibility and acceptability of the MRT design, as well as to compare acceptability and preliminary impact of two types of intervention messages in a sample of 65 postpartum mothers with histories of heavy episodic drinking.

The MRT was conducted using the Catalyst app, which was available for download on participants' personal smartphones. Participants completed ecological momentary assessment (EMA) surveys twice per day for 28 days. Following EMA completion, participants were randomized to receive a maternal-focused message (.40 probability), a drinking-focused message (.40 probability), or no message (.20 probability). If randomized to receive a message, participants would receive an intervention message that was selected at random from one of the 60 available messages in that condition, with each message having an equal probability of being selected. Following message receipt, participants were sent two questions asking whether the message was helpful (yes, no, not sure) and how the message made them feel (empowered, judged, understood, seen, confident, misunderstood, bad about myself, good, bad). Outcomes were assessed via EMA 15 minutes after delivery of the intervention message.

ELIGIBILITY:
Inclusion Criteria:

* adult women ages 18-45 years who gave birth to an infant that will remain in their care
* English-speaking
* own a text-enabled cell phone
* report a score of 2 or higher on the T-ACE alcohol risk screener AND (a) drinking weekly or more often in the past month OR (b) having 4 or more standard drinks at least monthly in the 12 months prior to becoming pregnant.

Exclusion Criteria:

* women age 46 years or older
* women who did not recently give birth to an infant
* women who gave birth to an infant but that infant is not in their care
* individuals who do not speak English
* women who report a score of less than 2 on the T-ACE alcohol risk screener
* women who do not report either weekly or more drinking in the past month OR having 4 or more standard drinks at least monthly in the 12 months prior to becoming pregnant.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Dauber, PhD, Principal Investigator — Partnership to End Addiction (formerly CASAColumbia)
Locations (1):
- Partnership to End Addiction, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We received 1408 valid eligibility screens, of which 1161 were complete. Of the 1161 completed eligibility screens, 771 participants met eligibility criteria for the study and 216 provided informed consent to participate. of the 216 participants who provided informed consent, 103 completed the baseline survey, 70 completed the training, and 66 enrolled in the study. One participant withdrew from the study shortly after enrolling, leaving a total sample size of 65.
Groups:
- Experimental: Text Messaging Intervention: The intervention consisted of text messages that were either maternal-focused (focused on the transition to motherhood) or drinking-focused (focused on reducing alcohol use). Each EMA survey (received twice daily) served as an intervention decision point. At each decision point, participants were randomized by the Catalyst app to receive a maternal message (.40 probability), a drinking message (.40 probability) or no message (.20 probability).
Period: Overall Study
Arm/Group | Experimental: Text Messaging Intervention
Started | 66
Completed | 65
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: We did not include the one participant who withdrew from the study in any analyses since she withdrew almost immediately after enrolling.
Arm/Group | Experimental: Text Messaging Intervention
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.26 (6.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 37
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: MRT Feasibility
Description: Proportion of EMA surveys completed out of total delivered.
Time Frame: Surveys were delivered 4 times per day (2 EMA, 2 proximal outcome surveys) on each of the 28 days of the intervention period.
Population: All participants who completed the study were included in the analysis of MRT feasibility.
Measure: Number; unit: percentage of surveys completed
Arm/Group | Experimental: Text Messaging Intervention
Number analyzed (Participants) | 65
percentage of surveys completed | 77.05

2. Primary Outcome: MRT Acceptability
Description: MRT acceptability was assessed via a 9-item scale assessing burden associated with the study. Cronbach's alpha in the sample was 0.88. Items were rated on a 1 to 7 scale, with higher scores reflecting higher burden. Scores on each item were averaged to create a total score ranging from 1 to 7. The average total score is reported.
Time Frame: Assessed on the final day of the 28-day MRT.
Population: All participants who completed the acceptability survey are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Text Messaging Intervention
Number analyzed (Participants) | 57
score on a scale | 2.31 (1.53)

3. Primary Outcome: Alcohol Use
Description: At each EMA survey/randomization decision point, participants were asked if they drank any alcohol in the prior hour (yes or no). At each proximal outcome survey (15 minutes after randomization), participants were asked if they drank any alcohol since their last survey (yes or no). The outcome is reported as the percent of participants who endorsed alcohol use on the proximal outcome survey, after randomization.
Time Frame: Assessed at each proximal outcome survey, twice per day for 28 days.
Population: All 65 participants are represented in each condition as each participant is randomized multiple times per day.
Measure: Number; unit: proximal outcome surveys
Units Other Than Participants: observations
Groups:
- Control/No Message: Randomized to receive no intervention message.
- Intervention Message (Drinking and Maternal Combined): Randomized to receive an intervention message--drinking and maternal focused messages combined.
- Maternal Focused Message: Randomized to receive a maternal focused message
- Drinking Focused Message: Randomized to receive a drinking focused message
Arm/Group | Control/No Message | Intervention Message (Drinking and Maternal Combined) | Maternal Focused Message | Drinking Focused Message
Number analyzed (Participants) | 65 | 65 | 65 | 65
Number analyzed (observations) | 411 | 1734 | 891 | 843
proximal outcome surveys | 16 | 58 | 31 | 27

4. Secondary Outcome: Maternal Self Efficacy
Description: At each proximal outcome survey, participants rated their confidence in their ability to meet their baby's needs over the next hour on a scale of 1 (not at all confident) to 7 (extremely confident). Higher numbers indicated greater maternal self-efficacy.
Time Frame: Assessed at each proximal outcome survey, twice per day for 28 days, regarding the next hour.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: observations
Arm/Group | Control/No Message | Intervention Message (Drinking and Maternal Combined) | Maternal Focused Message | Drinking Focused Message
Number analyzed (Participants) | 65 | 65 | 65 | 65
Number analyzed (observations) | 390 | 1655 | 847 | 808
score on a scale | 6.54 (0.93) | 6.57 (0.87) | 6.54 (0.89) | 6.61 (0.85)

5. Secondary Outcome: Drinking Self-Efficacy
Description: At each proximal outcome survey, participants rated their confidence in their ability to avoid drinking alcohol in the next hour on a scale of 1 (not at all confident) to 7 (extremely confident). Higher scores indicated higher drinking self-efficacy.
Time Frame: Assessed at each proximal outcome survey, twice per day for 28 days, regarding the next hour.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: observations
Arm/Group | Control/No Message | Intervention Message (Drinking and Maternal Combined) | Maternal Focused Message | Drinking Focused Message
Number analyzed (Participants) | 65 | 65 | 65 | 65
Number analyzed (observations) | 414 | 1742 | 895 | 847
score on a scale | 6.26 (1.34) | 6.37 (1.24) | 6.35 (1.24) | 6.39 (1.24)

6. Secondary Outcome: Motivation
Description: At each proximal outcome survey, participants were asked to rate how committed they are to not drink alcohol in the next hour on a scale of 1 (not at all committed) to 7 (extremely committed). Higher scores indicate higher motivation to avoid alcohol.
Time Frame: Assessed at each proximal outcome survey, twice a day for 28 days, regarding the next hour.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: observations
Arm/Group | Control/No Message | Intervention Message (Drinking and Maternal Combined) | Maternal Focused Message | Drinking Focused Message
Number analyzed (Participants) | 65 | 65 | 65 | 65
Number analyzed (observations) | 414 | 1743 | 896 | 847
score on a scale | 6.13 (1.52) | 6.21 (1.42) | 6.21 (1.39) | 6.20 (1.45)

7. Secondary Outcome: Urge to Drink
Description: At each proximal outcome survey, participants rated the extent of their urge to drink "right now" on a scale from 1 (very low) to 7 (very high). Higher scores indicate higher urge to drink alcohol.
Time Frame: Assessed at each proximal outcome survey, twice a day for 28 days.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: observations
Arm/Group | Control/No Message | Intervention Message (Drinking and Maternal Combined) | Maternal Focused Message | Drinking Focused Message
Number analyzed (Participants) | 65 | 65 | 65 | 65
Number analyzed (observations) | 413 | 1734 | 892 | 842
score on a scale | 1.94 (1.37) | 1.92 (1.31) | 1.96 (1.34) | 1.88 (1.29)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire 28 day MRT period.
Arm/Group | Experimental: Text Messaging Intervention
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT04719390/Prot_SAP_000.pdf